CLINICAL TRIAL: NCT03751111
Title: Treatment of Chronic Itch in Patients Under Arsenic Exposure With Sublingual Naloxone: A Double-blind Randomized Controlled Trial
Brief Title: Treatment of Chronic Itch in Patients Under Arsenic Exposure With Naloxone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Minxue Shen, Professor, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/NAL/CSU/PRU
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pruritus
Keywords: arsenic exposure; naloxone; placebo; single-blind randomized trial
MeSH Terms: interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two arms using a computer-generalized sequence of random numbers.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will not be informed whether the drug they received is naloxone or placebo. The investigators will remove the package of the drugs and use the unified package for both of the drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naloxone (Experimental): Naloxone at an sublingual dose of 0.4 mg daily will be given to each subject.
  Interventions: Drug: Naloxone
- Placebo (Placebo Comparator): Sublingual placebo will be given to each subject.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naloxone — Naloxone at an sublingual dose of 0.4 mg daily for one week will be given to each subject. Subjects will self-administer the drug at supervision in the primary care center.
  Arms: Naloxone
Drug: Placebo — Placebo will be given to each subject for one week. Subjects will self-administer the drug at supervision in the primary care center.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of sublingual naloxone in the treatment of chronic itch in patients under arsenic exposure.

DETAILED DESCRIPTION:
This study aims to determine the efficacy and safety of sublingual naloxone in the treatment of chronic, refractory itch in patients under long-term arsenic exposure. In this study, 120 subjects with a moderate-to-severe symptom of itching (numeric rating scale, NRS≥3) will be recruited and randomly treated with either sublingual naloxone (60 subjects) or placebo (60 subjects). The severity of itching will be evaluated in the wash out phase, baseline, and one week after the treatment through reporting of subjective symptomatology (itch NRS) via the interview. Quality of sleep measured by the Pittsburgh Sleep Quality Index (PSQI) and Dermatology Life Quality Index (DLQI) will serve as the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over and without diseases except arsenic-related pruritus
2. Ability to study protocol and to give informed consent by himself/herself voluntarily
3. The number of male or female subjects is required more than 1/3 of the total number of subjects
4. Numeric Rating Sscale≥3 at the baseline
5. Subjects taking hormone-containing medications must be on a stable dose for 6 months prior to study start to avoid any confounding influence on sensory and pain perception

Exclusion Criteria:

1. Use of oral anti-inflammatory medications for 2 weeks prior to the study start.
2. Use of oral anti-histamines for 2 weeks prior to the study start.
3. Use of topical or oral anti-pruritic agents for 2 weeks prior to the study start.
4. Use of oral neuromodulatory agents for 2 months prior to study start.
5. Current use of chronic pain medications (including opioids, antidepressants and anti-epileptic drugs).
6. Use of nicotine-containing products for the past 6 months prior to study start.
7. History of basic itchy dermatological diseases before such as eczema wich may influence the judgement of drug efficacy.
8. Unstable thyroid function within the past 6 months prior to study start to exclude thyroid-related neuropathy.
9. Known history of central or peripheral nervous system dysfunction.
10. History of acute hepatitis, chronic liver disease or end stage liver disease.
11. History of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome.
12. History of neuropathy associated with chronic obstructive pulmonary disease, diabetes mellitus, documented exposure to organophosphates or heavy metals or polychlorinated biphenyls.
13. Known nutritional deficiency (vitamin B12, vitamin D, iron or zinc) within 3 months prior to the study start.
14. Use of illicit drugs within the past 6 months prior to study start.
15. Lyme disease, porphyria, rheumatoid arthritis, Hansen's disease (leprosy) or use of antineoplastic chemotherapeutic agents.
16. Patients considered by researchers that are not suitable to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Xiao, Ph.D, Principal Investigator — Xiangya Hospital of Central South University; Minxue Shen, Ph.D, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol; Statistical Analysis Plan (SAP); Informed Consent Form (ICF) can be shared for the purpose of academic communication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the official start of the trial to the end of the trial
Access Criteria: Describe clearly about the reason of review

REFERENCES:
- [Background] Xiao Y, Huang X, Jing D, Huang Y, Zhang X, Shu Z, Huang Z, Su J, Li J, Zhang J, Chen M, Chen X, Shen M. Assessment of the Dermatology Life Quality Index (DLQI) in a homogeneous population under lifetime arsenic exposure. Qual Life Res. 2018 Dec;27(12):3209-3215. doi: 10.1007/s11136-018-1969-2. Epub 2018 Sep 10. PMID 30203303

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naloxone | Placebo
Started | 62 | 64
Completed | 50 | 32
Not Completed | 12 | 32
Not completed — Lack of Efficacy | 9 | 30
Not completed — Adverse Event | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naloxone | Placebo | Total
Number analyzed (Participants) | 62 | 64 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9) | 60 (9) | 59 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 35 | 38 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 62 | 64 | 126
Region of Enrollment [Number; unit: participants]
  China | 62 | 64 | 126
Numeric Rating Scale for Itch [Mean (Standard Deviation); unit: units on a scale] — Numeric Rating Scale (NRS) for Itch is a self-reported scale to measure the intensity of itch, with a range of score from 0 to 10. Higher scores indicate stronger itching, with a score of 1 or 2 suggesting mild itching, a score between 3 and 6 suggesting moderate itching, and a greater than 7 indicating severe itching.
  units on a scale | 8.18 (1.77) | 8.58 (1.56) | 8.38 (1.66)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale for Itch
Description: Participants will be invited to report the severity of itch using the Numeric Rating Scale (NRS) for Itch at the baseline and week 1 of the trial. Numeric Rating Scale (NRS) for Itch is a self-reported scale to measure the intensity of itch, with a range of score from 0 to 10. Higher scores indicate stronger itching, with a score of 1 or 2 suggesting mild itching, a score between 3 and 6 suggesting moderate itching, and a greater than 7 indicating severe itching.
Time Frame: 1 week
Population: Intention-to-treat population
Measure: Mean (Standard Deviation); unit: score on a scale (0~10)
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 62 | 64
score on a scale (0~10) | 6.42 (2.15) | 7.8 (1.99)

2. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: Measured by the Pittsburgh Sleep Quality Index (PSQI) at baseline and week 1 of the trial. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.
Time Frame: 1 week
Measure: Median (Inter-Quartile Range); unit: units on a scale (0-21)
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 62 | 64
units on a scale (0-21) | 9.5 [5 to 13] | 10.0 [6 to 12.5]

3. Secondary Outcome: Serological Indicator
Description: Level of serum beta-endorphin will be tested at baseline and week 1 of the trial
Time Frame: 1 week
Reporting Status: Not Posted

4. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: Dermatology Life Quality Index (DLQI) at baseline and week 1 of the trial. It consists of ten questions which ask about symptoms, feelings, daily activities, leisure, work, school, personal relationships, and treatment. Every question asked relates to the previous week. The user can tick a box in either: 'not at all', 'a little', 'a lot' or 'very much'. Questions are scored from 0 to 3 and totalled, giving an overall score out of 30. The final score ranges from 0 (no impact on quality of life) to 30 (maximum impairment).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale (0-30)
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 62 | 64
units on a scale (0-30) | 9.2 (6.7) | 12.1 (6.2)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Naloxone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 3/62 | 2/64
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naloxone (N=62) | Placebo (N=64)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03751111/Prot_SAP_000.pdf